CLINICAL TRIAL: NCT02505295
Title: Evaluation of Selenium Supplementation in Ischemic Stroke Outcome
Brief Title: Selenium and Ischemic Stroke Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant professor, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1421
Record Dates: First submitted 2015-07-11; First posted 2015-07-22 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Selenium; selenium-cisplatin conjugate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a feasibility/pilot study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- selenium (Active Comparator): vial selenium (selenase 500 microgr ) 2000 microgram stat and 1000 microgram daily for 5 days
  Interventions: Dietary Supplement: Selenium
- normal saline (Placebo Comparator): 40 cc normal saline stat and 20 cc daily for 5 days( in vials like selenase vial)
  Interventions: Drug: normal saline

INTERVENTIONS:
Dietary Supplement: Selenium — 4 vials selenase stat and 2 vials daily for 5 days
  Other Names: selenase; Selenium selenite
  Arms: selenium
Drug: normal saline — Normal saline infusion like intervention group
  Other Names: Sodium chloride 0.9%
  Arms: normal saline

SUMMARY:
Selenium is a trace element essential to human health.Selenium protection against cellular damage by oxygen radicals is accomplished through selenoproteins. Ischemic stroke is associated with the generation of oxygen free radicals resulting in a condition of oxidative stress. Supplementing stroke patients with antioxidant nutrients may improve survival.

ELIGIBILITY:
Inclusion Criteria:

1. Accepted ischemic stroke by brain CT or MRI during last 72 h
2. Ischemic stroke in Middle Cerebral Artery territory
3. Volume of stroke at list one third of MCA territory
4. written informed consent.

Exclusion Criteria:

1. Known allergy to selenium
2. Severe renal failure( cr clearance under 50 ml/min or serum cr upper than 2
3. Severe hepatic failure( total bill upper than 2 or ALT/AST 5 time upper than normal limit)
4. Severe neurodegenerative disease such as severe dementia, alzheimer and Parkinson
5. Pregnancy or lactation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale(NIHSS) | up to 3 days
  The primary outcome of interest in this study was defined as at least 25% reduction in NIHSS score in day 7 or at the discharge in selenium group compared with control; as an indicator of short term outcome.
modified Rankin Scale (MRS) | at day 5-8
  The primary outcome of interest in this study was defined as at least 1 point reduction in mRS score in day 7 or at the discharge in selenium group compared with control; as an indicator of short term outcome.

SECONDARY OUTCOMES:
Barthel index | 3 months after discharge
  The secondary outcome defined as Barthel index >75 three months after stroke, which indicates assisted independence, for long term outcome evaluation and comparison of mortality rate during the study follow-up between groups.

CONTACTS AND LOCATIONS:
Overall Officials: athena sharifi razavi, MD, Study Chair — assistant professor in neurology
Locations (1):
- Athena Sharifi Razavi, Sari, Mazandaran, Iran